CLINICAL TRIAL: NCT01208181
Title: A Phase III, Two-Part, Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial to Assess the Relative Efficacy and Tolerability of Two Doses of MK-0663/Etoricoxib in Patients With Rheumatoid Arthritis
Brief Title: A Two-Part, 12-Week Study of Etoricoxib as a Treatment for Rheumatoid Arthritis (RA) (MK-0663-107)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0663-107; 2010-019871-31 (EudraCT Number)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Etoricoxib 60 mg/Etoricoxib 60 mg (Experimental): The etoricoxib 60 mg/etoricoxib 60 mg treatment sequence will receive etoricoxib 60 mg tablets administered orally once daily for 6 weeks in Part 1 and Part 2 of the study.
  Interventions: Drug: Etoricoxib 60 mg; Drug: Placebo to Etoricoxib 60 mg
- Etoricoxib 60 mg/Etoricoxib 90 mg (Experimental): The etoricoxib 60 mg/etoricoxib 90 mg treatment sequence will receive etoricoxib 60 mg tablets administered orally once daily for 6 weeks in Part 1 and etoricoxib 90 mg tablets administered orally once daily for 6 weeks in Part 2 of the study.
  Interventions: Drug: Etoricoxib 60 mg; Drug: Placebo to Etoricoxib 60 mg
- Etoricoxib 90 mg (Experimental): The etoricoxib 90 mg treatment sequence will receive etoricoxib 90 mg tablets administered orally once daily for 6 weeks in Part 1 and will not participate in Part 2 of the study.
  Interventions: Drug: Etoricoxib 90 mg; Drug: Placebo to Etoricoxib 90 mg
- Placebo (Placebo Comparator): The placebo treatment sequence will receive matching placebo to etoricoxib tablets administered orally once daily for 6 weeks in Part 1 and will not participate in Part 2 of the study.
  Interventions: Drug: Placebo to Etoricoxib 60 mg; Drug: Placebo to Etoricoxib 90 mg

INTERVENTIONS:
Drug: Etoricoxib 60 mg — One tablet orally once daily for 6 weeks.
  Other Names: MK-0663
  Arms: Etoricoxib 60 mg/Etoricoxib 60 mg; Etoricoxib 60 mg/Etoricoxib 90 mg
Drug: Etoricoxib 90 mg — One tablet orally once daily for 6 weeks.
  Other Names: MK-0663
  Arms: Etoricoxib 90 mg
Drug: Placebo to Etoricoxib 60 mg — One tablet orally once daily for 6 weeks.
  Arms: Etoricoxib 60 mg/Etoricoxib 60 mg; Etoricoxib 60 mg/Etoricoxib 90 mg; Placebo
Drug: Placebo to Etoricoxib 90 mg — One tablet orally once daily for 6 weeks
  Arms: Etoricoxib 90 mg; Placebo

SUMMARY:
This is a 2-part (6 weeks duration for each part), randomized, double-blind, placebo-controlled study in participants with rheumatoid arthritis. The hypothesis is that etoricoxib (60 mg and 90 mg) administration will demonstrate superior efficacy compared to placebo after 6 weeks of treatment, as measured by the greater mean improvement from baseline in the Disease Activity Score C-Reactive Protein (DAS-28 CRP), and by the greater mean improvement in Patient Global Assessment of Pain (PGAP) from baseline over 6 weeks of treatment. Additionally, the added benefit of increasing the dose of etoricoxib from 60 mg to 90 mg will be assessed in the second part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 18 years of age in general good health (other than RA)
* Has an American College of Rheumatology Rheumatoid Clinical Response Criteria (ACR) Functional Class I, II, or III
* Has a diagnosis of RA at least 6 months ago and was at least 16 years of age when diagnosed
* Has a history of positive therapeutic benefit with nonsteroidal anti-inflammatory drugs (NSAIDs) and is taking an NSAID on a regular basis and at a therapeutic dose level and is not anticipated to undergo a change during the study

Exclusion Criteria:

* Has a concurrent medical/arthritic disease that could confound or interfere with evaluation of efficacy
* Has a history of gastric or biliary surgery (including gastric bypass surgery) or small intestine surgery that causes clinical malabsorption
* Has an active peptic (gastric or duodenal) ulcer or history of inflammatory bowel disease
* Has a confirmed medical diagnosis of ischemic heart disease, cerebrovascular disease, or peripheral artery occlusive disease
* Class II-IV congestive heart failure
* Has uncontrolled hypertension (systolic >160 mm Hg or diastolic > 90 mm Hg) at Visit 1 or Visit 2
* Has a clinical diagnosis of hepatic insufficiency defined as Child-Pugh score ≥5
* Has estimated glomerular filtration rate ≤30 mL/min
* Has a history of neoplastic disease within 5 years (exceptions: basal cell carcinoma or carcinoma in situ of the cervix)
* Is allergic to etoricoxib; history of a significant clinical or laboratory adverse experience associated with etoricoxib; hypersensitivity to aspirin or NSAIDs; or allergy to acetaminophen/paracetamol
* Has a personal or family history of an inherited or acquired bleeding disorder
* Requires oral corticosteroid therapy in excess of the equivalent of 10 mg daily of prednisone and/or have not been on a stable dose for at least 4 weeks prior to Visit 1 and/or whose dose is not expected to remain stable during the study
* Treated with B-cell depleting therapies within the past 6 months or anticipate this treatment during this trial
* Is a recreational or illicit drug use, or history within 5 years of drug or alcohol abuse/dependence;
* Is morbidly obese (defined as body mass index ≥40 kg/m^2)
* Is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1404 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2014-06-09 (Actual); Study Completion 2014-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bickham K, Kivitz AJ, Mehta A, Frontera N, Shah S, Stryszak P, Popmihajlov Z, Peloso PM. Evaluation of two doses of etoricoxib, a COX-2 selective non-steroidal anti-inflammatory drug (NSAID), in the treatment of Rheumatoid Arthritis in a double-blind, randomized controlled trial. BMC Musculoskelet Disord. 2016 Aug 8;17:331. doi: 10.1186/s12891-016-1170-0. PMID 27502582

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoricoxib 60 mg: The etoricoxib 60 mg treatment group received etoricoxib tablets 60 mg administered orally once daily in Part 1 of the study.
- Etoricoxib 90 mg: The etoricoxib 90 mg treatment sequence received etoricoxib tablets 90 mg administered orally once daily in Part 1 of the study.
- Etoricoxib 60 mg/Etoricoxib 60 mg: The etoricoxib 60 mg/etoricoxib 60 mg treatment sequence received etoricoxib tablets 60 mg administered orally once daily in Part 1 and Part 2 of the study.
- Etoricoxib 60/Etoricoxib 90mg: The etoricoxib 60 mg/etoricoxib 90 mg treatment sequence received etoricoxib tablets 60 mg administered orally once daily in Part 1 of the study and etoricoxib tablets 90 mg administered orally once daily in Part 2 of the study.
- Placebo: The placebo treatment group received placebo to etoricoxib tablets administered orally once daily in Part 1 of the study.
Period: Part 1
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Etoricoxib 60 mg/Etoricoxib 60 mg | Etoricoxib 60/Etoricoxib 90mg | Placebo
Started | 818 | 468 | 0 | 0 | 118
Completed | 719 (Six participants from this arm did not continue into Part II of the study) | 413 (Per protocol, participants in this arm did not continue into Part II of the study) | 0 | 0 | 96 (Per protocol, participants in this arm did not continue into Part II of the study)
Not Completed | 99 | 55 | 0 | 0 | 22
Not completed — Withdrawal by Subject | 11 | 10 | 0 | 0 | 0
Not completed — Technical problem | 5 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 10 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 3 | 0 | 0 | 1
Not completed — Lack of Efficacy | 37 | 12 | 0 | 0 | 17
Not completed — Adverse Event | 26 | 24 | 0 | 0 | 4
Period: Part 2
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Etoricoxib 60 mg/Etoricoxib 60 mg | Etoricoxib 60/Etoricoxib 90mg | Placebo
Started | 0 (Per protocol, there were no participants in this arm during Part II of the study) | 0 (Per protocol, there were no participants in this arm during Part II of the study) | 350 (Participants receiving etoricoxib 60 mg in Part I received etoricoxib 60 mg in Part II of the study) | 363 (Participants receiving etoricoxib 60 mg in Part I received etoricoxib 90 mg in Part II of the study) | 0 (Per protocol, participants did not receive placebo during Part II of the study)
Completed | 0 | 0 | 334 | 343 | 0
Not Completed | 0 | 0 | 16 | 20 | 0
Not completed — Adverse Event | 0 | 0 | 6 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 5 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Placebo | Total
Number analyzed (Participants) | 818 | 468 | 118 | 1404
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (11.9) | 54.0 (12.3) | 53.6 (11.0) | 53.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 677 | 395 | 100 | 1172
  Male | 141 | 73 | 18 | 232
Disease Activity Score using C reactive protein (DAS28-CRP) [Mean (Standard Deviation); unit: Scores on a scale] — The DAS28-CRP index (0 - 10 Range) is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity, and C-reactive protein (CRP). For each observation (Baseline, Week 2, 4, 6, 10, 12), components were combined into a single DAS28-CRP score using the following algorithm: 0.56*square root (sqrt) (tender joint count [28])+0.28*sqrt(swollen joint count [28] )+0.36* ln(crp+1) + 0.014* Patient Global Assessment of Disease Activity + 0.96. (N = 732, 426, 103 for Etoricoxib 60 mg, Etoricoxib 90 mg, and Placebo).
  Scores on a scale | 5.64 (0.99) | 5.62 (1.00) | 5.65 (1.12) | 5.63 (1.00)
Patient Global Assessment of Pain [Mean (Standard Deviation); unit: Scores on a scale] — A participant overall assessment of pain on a visual analog scale (VAS) were assessed with a question concerning the amount of pain due to arthritis during the past 48 hours. Pain was assessed on an 100 mm VAS scale with a left-hand marker "no pain" (0 mm) or right-hand marker "extreme pain" (100 mm). (N = 751, 430, 108 for Etoricoxib 60 mg, Etoricoxib 90 mg, and Placebo)
  Scores on a scale | 70.84 (15.50) | 70.58 (15.02) | 74.08 (14.23) | 71.02 (15.24)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change From Baseline in DAS28-CRP in Part 1 (Etoricoxib vs. Placebo)
Description: Disease Activity Score Using C-Reactive Protein [DAS28-CRP] (0 - 10 Range). The DAS28-CRP index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity, and C-reactive protein (CRP). For each observation (Baseline, Week 2, 4, 6, 10, 12), components were combined into a single DAS28-CRP score using the following algorithm: 0.56*square root (sqrt) (tender joint count [28])+0.28*sqrt(swollen joint count [28] )+0.36* ln(crp+1) + 0.014* Patient Global Assessment of Disease Activity + 0.96. The primary objectives of the study compared the efficacy of etoricoxib (90 mg, 60 mg) to placebo in Part 1 of this study so data for only these 3 arms are displayed.
Time Frame: Baseline and Week 6
Population: The modified intention-to-treat (mITT) population in Part 1 consisted of all randomized participants receiving at least 1 dose of study medication, had baseline data for the analysis endpoint, and least one post-randomization measurement for the analysis endpoint that was collected within 3 days after the last dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Placebo
Number analyzed (Participants) | 732 | 426 | 103
Scores on a scale | -1.39 [-1.48 to -1.30] | -1.37 [-1.48 to -1.26] | -1.10 [-1.29 to -0.90]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Tukey-Ciminera-Heysetrend test; Difference in least squares mean = -0.29, 95% CI 2-sided [-0.49 to -0.09]
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority or Other; p = 0.034, Tukey-Ciminera-Heysetrend test; Difference in least squares mean = -0.27, 95% CI 2-sided [-0.48 to -0.06]

2. Primary Outcome: Time-Weighted Average Change From Baseline in Patient Global Assessment of Pain in Part 1 (Etoricoxib vs. Placebo)
Description: A participant overall assessment of pain on a visual analog scale (VAS) was assessed with a question concerning the amount of pain due to arthritis during the past 48 hours. Pain was assessed on an 100 mm VAS scale with a left-hand marker "no pain" (0 mm) or right-hand marker "extreme pain" (100 mm). The primary objectives of the study compared the efficacy of etoricoxib (90 mg, 60 mg) to placebo in Part 1 of this study so data for only these 3 arms are displayed.
Time Frame: Baseline and Week 6
Population: The mITT population in Part 1 consisted of all randomized participants receiving at least 1 dose of study medication, had baseline data for the analysis endpoint, and least one post-randomization measurement for the analysis endpoint that was collected within 3 days after the last dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Placebo
Number analyzed (Participants) | 751 | 430 | 108
Scores on a scale | -28.25 [-30.05 to -26.44] | -30.96 [-33.13 to -28.79] | -20.26 [-24.04 to -16.48]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Tukey-Ciminera-Heyse trend test; Difference in least squares mean = -7.99, 95% CI 2-sided [-11.85 to -4.13]
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Tukey-Ciminera-Heyse trend test; Difference in least squares mean = -10.70, 95% CI 2-sided [-14.74 to -6.66]

3. Secondary Outcome: Time-Weighted Average Change From Baseline in DAS28-CRP in Part 1 (Etoricoxib 90 mg vs. Etoricoxib 60 mg)
Description: Disease Activity Score Using C-Reactive Protein [DAS28-CRP] (0 - 10 Range). The DAS28-CRP index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity, and C-reactive protein (CRP). For each observation (Baseline, Week 2, 4, 6, 10, 12), components were combined into a single DAS28-CRP score using the following algorithm: 0.56*square root (sqrt) (tender joint count [28])+0.28*sqrt(swollen joint count [28] )+0.36* ln(crp+1) + 0.014* Patient Global Assessment of Disease Activity + 0.96. The key secondary objectives compared the relative efficacy between etoricoxib 90 mg and 60 mg in Part 1 of this study so data for only these 2 arms are displayed.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 732 | 426
Scores on a scale | -1.39 [-1.48 to -1.30] | -1.37 [-1.48 to -1.26]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p = 0.730, Tukey-Ciminera-Heysetrend test; Difference in least squares mean = 0.02, 95% CI 2-sided [-0.10 to 0.14]

4. Secondary Outcome: Time-Weighted Average Change From Baseline in Patient Global Assessment of Pain in Part 1 (Etoricoxib 90 mg vs. Etoricoxib 60 mg)
Description: A participant overall assessment of pain on a visual analog scale (VAS) was assessed with a question concerning the amount of pain due to arthritis during the past 48 hours. Pain was assessed on an 100 mm VAS scale with a left-hand marker "no pain" (0 mm) or right-hand marker "extreme pain" (100 mm). The key secondary objectives compared the relative efficacy between etoricoxib 90 mg and 60 mg in Part 1 of this study so data for only these 2 arms are displayed.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 751 | 430
Scores on a scale | -28.25 [-30.05 to -26.44] | -30.96 [-33.13 to -28.79]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p = 0.019, Tukey-Ciminera-Heyse trend test; Difference in least squares mean = -2.71, 95% CI 2-sided [-4.98 to -0.45]

5. Secondary Outcome: Average Change From Week 6 in Patient Global Assessment of Pain Over Weeks 10 and 12 in Part 2 Among Pain Inadequate Responders From Part 1
Description: A participant overall assessment of pain on a visual analog scale (VAS) was assessed with a question concerning the amount of pain due to arthritis during the past 48 hours. Pain was assessed on an 100 mm VAS scale with a left-hand marker "no pain" (0 mm) or right-hand marker "extreme pain" (100 mm). In those participants who were considered inadequate responders to etoricoxib 60 mg in Part 1 (defined as a participant with <50% improvement from baseline in PGAP [VAS] at Week 6), the incremental benefit of increasing the etoricoxib dose from 60 mg (in Part 1) to 90 mg (in Part 2) compared to remaining on 60 mg in Part 2 was evaluated via average change from Week 6 over Weeks 10 and 12 in Patient Global Assessment of Pain score. Therefore, data for only these 2 arms are displayed.
Time Frame: Week 6 and Week 10 to Week 12
Population: This population (a subpopulation of the mITT population) was composed of pain inadequate responder (PIRs) in Part 1. PIRs were defined as participants with <50% improvement from baseline in Patient Global Assessment of Pain (VAS) at Week 6 and received at least one dose of study medication in Part 2.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Etoricoxib 60 mg/Etoricoxib 60 mg: The etoricoxib 60 mg/etoricoxib 60 mg treatment sequence will receive etoricoxib 60 mg tablets administered orally once daily in Part 1 and Part 2 of the study.
- Etoricoxib 60 mg/Etoricoxib 90 mg: The etoricoxib 60 mg/etoricoxib 90 mg treatment sequence will receive etoricoxib 60 mg tablets administered orally once daily in Part 1 and etoricoxib 90 mg tablets Part 2 of the study.
Arm/Group | Etoricoxib 60 mg/Etoricoxib 60 mg | Etoricoxib 60 mg/Etoricoxib 90 mg
Number analyzed (Participants) | 188 | 187
Scores on a scale | -11.96 [-14.96 to -8.97] | -10.35 [-13.32 to -7.39]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg/Etoricoxib 60 mg vs Etoricoxib 60 mg/Etoricoxib 90 mg; Test type: Superiority or Other; p = 0.327, covariance model; Difference in the least squares mean = 1.61, 80% CI 2-sided [-0.49 to 3.71]

6. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to 112 days
Population: All Subjects as Treated (ASaT) population, defined as all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the ASaT population.
Measure: Number; unit: Percentage of participants
Groups:
- Etoricoxib 60 mg - Part 1: The etoricoxib 60 mg treatment group received etoricoxib tablets 60 mg administered orally once daily in Part 1 of the study.
- Etoricoxib 90 mg - Part 1: The etoricoxib 90 mg treatment sequence received etoricoxib tablets 90 mg administered orally once daily in Part 1 of the study.
- Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2: The etoricoxib 60 mg/etoricoxib 60 mg treatment sequence will receive etoricoxib tablets 60 mg administered orally once daily in Part 1 and Part 2 of the study.
- Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2: The etoricoxib 60 mg/etoricoxib 90 mg treatment sequence will receive etoricoxib tablets 60 mg administered orally once daily in Part 1 of the study and etoricoxib tablets 90 mg administered orally once daily in Part 2 of the study.
- Placebo - Part 1: The placebo treatment group received placebo to etoricoxib tablets administered orally once daily in Part 1 of the study.
Arm/Group | Etoricoxib 60 mg - Part 1 | Etoricoxib 90 mg - Part 1 | Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2 | Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2 | Placebo - Part 1
Number analyzed (Participants) | 819 | 467 | 350 | 363 | 118
Percentage of participants | 30.3 | 36.0 | 19.1 | 24.5 | 25.4

7. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 6
Time Frame: Up to Week 12
Population: ASaT population defined as all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the ASaT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Etoricoxib 60 mg - Part 1 | Etoricoxib 90 mg - Part 1 | Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2 | Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2 | Placebo - Part 1
Number analyzed (Participants) | 819 | 467 | 350 | 363 | 118
Percentage of participants | 3.3 | 5.1 | 1.4 | 1.9 | 3.4

ADVERSE EVENTS:
Time Frame: Up to 112 days
Description: The All Participants as Treated (APaT) population was used for the analysis of safety data in this study and consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Arm/Group | Etoricoxib 60 mg - Part 1 | Etoricoxib 90 mg - Part 1 | Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2 | Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2 | Placebo - Part 1
Serious Adverse Events (participants affected / at risk) | 7/819 | 2/467 | 4/350 | 5/363 | 0/118
Other Adverse Events (participants affected / at risk) | 25/819 | 17/467 | 6/350 | 6/363 | 6/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 60 mg - Part 1 (N=819) | Etoricoxib 90 mg - Part 1 (N=467) | Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2 (N=350) | Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2 (N=363) | Placebo - Part 1 (N=118)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 60 mg - Part 1 (N=819) | Etoricoxib 90 mg - Part 1 (N=467) | Etoricoxib 60mg/Etoricoxib 60mg - Part 1/2 (N=350) | Etoricoxib 60mg/Etoricoxib 90mg - Part 1/2 (N=363) | Placebo - Part 1 (N=118)
Headache (Nervous system disorders) | 25 (27) | 17 (27) | 6 (6) | 6 (7) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.